CLINICAL TRIAL: NCT06139484
Title: Stanford Neuromodulation Therapy (SNT) for Non-suicidal Self-injury (NSSI)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Head, Dept of Neurology & Medical Psychology, Director, Cognitive Neuropsychology Lab, PRC, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHMU-SNT-NSSI
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Transcranial Magnetic Stimulation; Non-suicidal Self-injury
Keywords: Transcranial Magnetic Stimulation; Non-suicidal Self-injury
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SNT Group (Active Comparator): Patients will be treated with neuronavigated transcranial magnetic stimulation. The treatment protocol is 90% motor threshold (RMT) stimulation intensity for 60 cycles of 10 triplet pulses each at a frequency of 50 Hz, in 2-second stimulation sequences (5 Hz) with 8-second intervals. Stimulation treatments were performed hourly. Ten treatments per day (18,000 pulses/day) for 5 consecutive days (90,000 pulses total).
  Interventions: Device: Transcranial Magnetic Stimulation
- rTMS Group (Other): Patients will be treated with the normal non-neuronavigated transcranial magnetic stimulation. The treatment protocol is 90%-100% RMT stimulation intensity; 10 Hz frequency for 4 seconds with 26 seconds of rest; 4,000 pulses per session; total duration 50 minutes, twice daily (8,000 pulses/day) for 5 days (40,000 pulses total).
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — The stimulations were performed by Magstim RAPID.

SUMMARY:
To investigate the treatment effect of Stanford Neuromodulation Therapy (SNT) on patients with Non-suicidal Self-injury (NSSI) and the underlying neural mechanism.

DETAILED DESCRIPTION:
This was a open-label clinical trial to assess the efficacy and underlying neural mechanism of SNT among patients with NSSI.

80 patients with NSSI diagnosed by DSM-5 were recruited from the Second Hospital of Anhui Medical University. After meeting the inclusion criteria and obtaining informed consent, All the participants were randomized (1:1) into two groups: SNT group and rTMS group.

Before the treatment, the Adolescent Non-suicidal Self-injury Assessment Questionnaire (ANSAQ) was obtained by a trained investigator to assess baseline severity. The patients had receiving a battery measure of neuropsychological tests(Hamilton depression/anxiety scale, Health Questionnaire-15) and magnetic resonance imaging (MRI) scan in multimodalities.

For SNT group, the treatment was performed once a day for 5 consecutive days. A Brainsight neuronavigation system was used to position the TMS coil over the individualized stimulation target at each session. Ten sessions of iTBS were delivered daily, for a total of 18,000 pulses per day. Stimulation was delivered at 90% of resting motor threshold (rMT).

For rTMS group, the treatment was also performed once a day for 5 consecutive days. Two sessions of rTMS were delivered daily. Each rTMS session comprised 100 trains of 4s duration at 10 Hz with inter-train intervals of 26 s (i.e., 4000 pulses per session). Stimulation was delivered at 90% of rMT.

In the second day after the last treatment, all the tests and MRI were reassessed. Patients were instructed to focus their answers on the past 1 week.

The clinical symptom and cognition of participants were followed in one week and one month after the last treatment.

ELIGIBILITY:
Inclusion Criteria:

* the patients were diagnosed by 2 or more senior clinical psychiatrists, meeting DSM-V criteria, and having 1 or more non-suicidal self-injurious behaviors in the last 6 months
* 12-18 years of age
* The medicine has not changed in the 4 weeks prior to or after this study, and if it has to be changed, the treatment medication is required to be at a subtherapeutic dosage level

Exclusion Criteria:

* the patients has suicidal ideation, or have committed suicidal behavior
* T1 or T2 weighted phase magnetic resonance images show focal brain lesions
* patients had neurological disorders such as epilepsy, or serious physical illnesses
* patients had history of substance abuse and drug dependence in the last 6 months or use of anticonvulsant drugs in the last 3 months
* patiens had received radial cranial electrical stimulation or magnetic stimulation treatment in the last 3 months, or received electroconvulsive therapy in the last 6 months
* patients had previous significant head trauma or with EEG abnormality in the last 1 month
* body-mounted devices unsuitable for treatment, such as pacemakers, artificial valves and other metal implants.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Adolescent Non-suicidalself-injury Assessment Questionnaire | baseline, the second day(immediately after the intervention),the seventh day(immediately after the intervention)
  The questionnaire consisted of 2 dimensions and 12 items, with 5 options for each item, namely, "none, occasional, sometimes, often and always", and was scored on a 5-point Likert scale from 0 to 4. The score for each item was summed up as the total score of the questionnaire, and the total mean score was divided by the number of items. The total mean score was divided by the number of items, and the higher the total mean score, the more serious the patients' non-suicidal Likert 5 self-injurious behaviors were.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HAMD) Score | baseline, the second day(immediately after the intervention),the seventh day(immediately after the intervention)
  The HAMD is a clinician-administered depression assessment and consists of 17 items with a total score range from 0 to 54. A higher score indicates a worse outcome.
Hamilton Anxiety Scale (HAMA) Score | baseline, the second day(immediately after the intervention),the seventh day(immediately after the intervention)
  The HAMA is a 14-item scale to measure the severity of anxiety symptoms, where each item is rated on a scale from 0 to 4. The HAMA total score ranges from 0 to 56, with lower scores indicating less anxiety symptoms.
Patient Health Questionnaire-15 (PHQ-15) scale | baseline, the second day(immediately after the intervention),the seventh day(immediately after the intervention)
  The PHQ-15 is a 15-item scale to measure the severity of somatic symptoms, where each item is rated on a scale from 0 to 2. The PHQ-15 total score ranges from 0 to 30, with lower scores indicating less somatic symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Yanghua Tian, PhD, Study Chair — Anhui Medical University
Locations (1):
- Anhui Medical University, Hefei, China